CLINICAL TRIAL: NCT01457456
Title: Biomarker for Morquio Disease AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Biomarker for Morquio Disease (BioMorquio)
Acronym: BioMorquio
Status: Withdrawn | Type: Observational
Why Stopped: Transition to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BM 06-2018
Record Dates: First submitted 2011-10-21; First posted 2011-10-24 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Morquio Syndrome; Accumulation of Mucopolysaccharides; Morquio Syndrome A; Morquio B Disease
Keywords: Biomarker; Morquio Disease
MeSH Terms: conditions — Mucopolysaccharidosis IV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of mass-spectometry 10 ml EDTA blood and a dry blood spot filter card are used. To prove the correct Morquio diagnosis in those patients where up to the enrollment in the study no genetic testing has been done, sequencing of Morquio will be done as routine diagnostic sequencing.
  The analyses will done in the Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Morquio disease

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Morquio disease from plasma

DETAILED DESCRIPTION:
Morquio syndrome (mucopolysaccharidosis type IV; MPS IV) is a mucopolysaccharide storage disease that exists in two forms (Morquio syndromes A and B) and occurs because of a deficiency of the enzymes N-acetyl-galactosamine-6-sulfatase and beta-galactosidase, respectively. A deficiency of either enzyme leads to the accumulation of mucopolysaccharides in the body, abnormal skeletal development, and additional symptoms. In most cases, individuals with Morquio syndrome have normal intelligence. The clinical features of MPS IV-B are less severe than those associated with MPS IV-A. Symptoms may include growth retardation, a prominent lower face, an abnormally short neck, knees that are abnormally close together (knock knees or genu valgum), flat feet, abnormal sideways and front-to-back or side-to-side curvature of the spine (kyphoscoliosis), abnormal development of the growing ends of the long bones (epiphyses) resulting in dwarfism, and/or a prominent breast bone (pectus carinatum) as well as bell shaped chest. Though the CNS and peripheral nerves are primarily not affected the bone defects may result in neurological symptoms such as spinal cord compression. Hearing loss, weakness of the legs, and/or additional abnormalities may also occur.

The mucopolysaccharidoses (MPS) are a group of inherited lysosomal storage disorders. Lysosomes function as the primary digestive units within cells. Enzymes within lysosomes break down or digest particular nutrients, such as certain carbohydrates and fats. In individuals with MPS disorders, deficiency or malfunction of specific lysosomal enzymes lead to an abnormal accumulation of certain complex carbohydrates (mucopolysaccharides or glycosaminoglycans) in the arteries, skeleton, eyes, joints, ears, skin and/or teeth. These accumulations may also be found in the respiratory system, liver, spleen, central nervous system, blood, and bone marrow. This accumulation eventually causes progressive damage to cells, tissues, and various organ systems of the body. There are several different types and subtypes of mucopolysaccharidosis. These disorders, with one exception, are inherited as autosomal recessive traits and all vary in their clinical phenotype. Within our clinical trial we focus on MPS type IV.

New methods, like mass-spectrometry give a good chance to characterize in the blood (plasma) of affected patents specific metabolic alterations that allow to diagnose in the future the disease earlier, with a higher sensitivity and specificity. Therefore it is the goal of the study to develop new biochemical markers from the plasma of the affected patients helping to benefit the patient by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

* Informed consent will be obtained from the patient or the parents before any study related procedures
* Patients older than 12 months
* The patient has a diagnosis of Morquio disease

EXCLUSION CRITERIA:

* No Informed consent from the patient or the parents before any study related procedures.
* Patients younger than 12 months
* The patient has no diagnosis of Morquio disease

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Morquio disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Morquio disease from blood (plasma) | 24 month
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker | 36 months
  the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (5):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka